CLINICAL TRIAL: NCT01428297
Title: A First-In-human Study to Evaluate Safety and Tolerability of Topical BPR277 in Healthy Volunteers, and Proof of Concept (PoC) Studies to Evaluate the Safety, Tolerability, and Efficacy of Topical BPR277 in Patients With Atopic Dermatitis and Netherton Syndrome
Brief Title: A Study Evaluating the Safety and Efficacy of Topical BPR277 for the Treatment of Atopic Dermatitis and Netherton Syndrome
Acronym: 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Clinical Disclosure Office, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CBPR277X2101; 2011-000917-38
Record Dates: First submitted 2011-08-19; First posted 2011-09-02 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2015-02

CONDITIONS: Healthy Volunteers; Atopic Dermatitis; Netherton Syndrome
Keywords: Atopic dermatitis; Eczema; Skin Diseases, Eczematous; Netherton syndrome; Skin Diseases, Genetic; BPR277
MeSH Terms: conditions — Dermatitis, Atopic; Netherton Syndrome; Eczema; Skin Diseases, Eczematous; Skin Diseases, Genetic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Cohort A and B, BPR277 and Placebo (vehicle) (Experimental)
  Interventions: Drug: BPR277 ointment (controlled application); Drug: Placebo (Vehicle)
- Part 2 BPR277 (Experimental)
  Interventions: Drug: BPR277 ointment
- Part 2 Placebo (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo (Vehicle)
- Part 3 BPR277 and Placebo (vehicle) (Experimental)
  Interventions: Drug: BPR277; Drug: Placebo (Vehicle)

INTERVENTIONS:
Drug: BPR277 ointment (controlled application)
  Arms: Cohort A and B, BPR277 and Placebo (vehicle)
Drug: Placebo (Vehicle)
  Arms: Cohort A and B, BPR277 and Placebo (vehicle)
Drug: BPR277 ointment
  Arms: Part 2 BPR277
Drug: Placebo (Vehicle)
  Arms: Part 2 Placebo (vehicle)
Drug: BPR277
  Arms: Part 3 BPR277 and Placebo (vehicle)
Drug: Placebo (Vehicle)
  Arms: Part 3 BPR277 and Placebo (vehicle)

SUMMARY:
The study is divided in 3 parts, starting with the safety assessment of BPR277 ointment in Healthy volunteers (Part 1). If found to be well tolerated in Part 1, BPR277 ointment will be assessed in two different patients groups to evaluate safety and efficacy in atopic dermatitis (Part 2) and in Netherton syndrome (Part 3).

ELIGIBILITY:
Inclusion Criteria:

Part 1 Healthy volunteers

* Healthy male and female subjects of non childbearing potential, 18 to 65 years of age inclusive and in good health

Part 2 Patients with atopic dermatitis:

* Male and female subjects, 18 to 65 years of age inclusive and having passed screening examinations
* Presence of atopic dermatitis confirmed by Itchy skin condition in the past 12 months (must have) Plus three or more of the following:

  1. History of involvement of the skin creases
  2. Personal history of asthma or hay fever
  3. History of generally dry skin in the past year
  4. Onset before age of 2 years
  5. Visible flexural dermatitis
* Diagnosis of at least moderate atopic dermatitis by the IGA and a minimum target area (right or left) situated on the forearm including the antecubital fossa with a corresponding baseline total lesional sign score (TLSS)

Part 3 Patients with Netherton Syndrome:

* Patients with Netherton syndrome, male and female subjects, 18 to 65 years of age inclusive and having passed screening examinations
* Confirmed diagnosis of Netherton syndrome (SPINK5 mutation or LEKTI deficiency in the skin).
* Minimum total lesional sign score NS (TLSS-NS) of 5-9 for two selected target areas at baseline. The TLSS-NS values need to be similar between the two areas at baseline.

Exclusion Criteria:

Part 1 Healthy volunteers :

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes or history of serious allergic reaction.
* Use of any prescription drugs, herbal supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing.

Part 2 Patients with atopic dermatitis:

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes or history of serious allergic reaction.
* History of abnormal skin reactivity to UV light. Unusual exposure to UV light in the previous 3 weeks to study start (screening), including tanning and sun beds.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential must use highly effective contraception (as further defined in study protocol)
* Use of topical prescription treatment for eczema within 1 week prior to initial dosing of topical corticosteroids (TCS).
* Recent previous treatment with systemic treatment including phototherapy. A washout period will be required for such patients to be eligible to participate in the trial.

Part 3 Patients with Netherton Syndrome:

* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes or history of serious allergic reaction.
* History of abnormal skin reactivity to UV light. Unusual exposure to UV light in the previous 3 weeks to study start (screening), including tanning and sun beds.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential must use highly effective contraception (as further defined in study protocol)
* Use of topical prescription treatment within 2 week prior to initial dosing of study drug.
* Recent previous treatment with systemic treatment. A washout period will be required for such patients to be eligible to participate in the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Systemic and local tolerability of BPR277 ointment, as measured by change in local tolerability score, number of adverse events and clinically significant changes in standard hematology, blood chemistry. | 2-4 weeks
Part 2 and 3: Patients with Atopic Dermatitis / Netherton syndrome: Change in Total Lesional Signs Score at the treated skin area | 4 weeks

SECONDARY OUTCOMES:
Part 2 and 3: Patients with Atopic Dermatitis / Netherton syndrome: Change for each sign comprising the total lesional signs score at the treated skin area | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (3):
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Fargo, North Dakota
- Novartis Investigative Site, Utrecht, The Netherlands, Netherlands

REFERENCES:
- See also: Results for CBPR277X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13551